CLINICAL TRIAL: NCT05083052
Title: Propolis in Reducing Dentin Hypersensitivity: a Randomized Clinical Trial
Brief Title: Propolis in Reducing Dentin Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Para (Other)
Responsible Party: Principal Investigator, Cecy Martins Silva, Clinical professor, Universidade Federal do Para
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UFPa - 0011
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Dentin Sensitivity
Keywords: Dentin Desensitizing Agents; Propolis.
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PLACEBO (Placebo Comparator): Carbonato de cálcio: 40,0%, Glicerina: 20,0%, Lauril Sulfato de sódio: 1,2%, Carboximetilcelulose: 2,0%, Goma xantana: 1,0%, Metilparabeno (nipagim): 0,15%, EDTA: 0,5%, Sacarina: 0,1%, Flavorizante: 0,75%, Água deionizada q.s.p - 100mL.
  Interventions: Other: Placebo
- PROPOLIS 10% (Experimental): Carbonato de cálcio: 40,0%, Glicerina: 20,0%, Lauril Sulfato de sódio: 1,2%, Carboximetilcelulose: 2,0%, Goma xantana: 1,0%, Metilparabeno (nipagim): 0,15%, EDTA: 0,5%, Sacarina: 0,1%, Flavorizante: 0,75%, Própolis a 10%, Água deionizada q.s.p - 100mL.
  Interventions: Other: Propolis 10%
- PROPOLIS 15% (Experimental): Carbonato de cálcio: 40,0%, Glicerina: 20,0%, Lauril Sulfato de sódio: 1,2%, Carboximetilcelulose: 2,0%, Goma xantana: 1,0%, Metilparabeno (nipagim): 0,15%, EDTA: 0,5%, Sacarina: 0,1%, Flavorizante: 0,75%, Própolis a 15%, Água deionizada q.s.p - 100mL.
  Interventions: Other: Propolis 15%

INTERVENTIONS:
Other: Propolis 15% — oothpaste formulation with 15% propolis.
  Arms: PROPOLIS 15%
Other: Propolis 10% — Toothpaste formulation with 10% propolis.
  Arms: PROPOLIS 10%
Other: Placebo — Formulation of toothpaste without active ingredient.
  Arms: PLACEBO

SUMMARY:
Objective: This randomized, double-blind, parallel, placebo-controlled clinical trial aims to evaluate the effect of propolis with two distinct concentrations (10% and 15%), and the impact on volunteers' quality of life.

Materials and methods: Volunteers meeting the inclusion and exclusion criteria will be randomized and allocated into three groups: Group 1- placebo - toothpaste without active ingredient, Group 2- toothpaste with 10% propolis and Group 3. - toothpaste with 15% propolis. Number of teeth will be used as sample unit, totaling 22 teeth per group. Volunteers will receive oral hygiene instruction with guidance to brush their teeth three times a day with toothpaste corresponding to the groups in which they will be allocated for 30 days. The evaluation of dentin hypersensitivity will be performed with three (3) evaluation times: baseline (immediately before the beginning of treatment), 15 and 30 days, through tactile and evaporative stimuli, using the visual analog scale (VAS). The self-reported evaluation of the volunteers will be done through a questionnaire before the beginning and after one month with the completion of the research to determine the impact of treatment on their quality of life. The data regarding HD in VAS, if present normal distribution, will be used Two-way analysis of variance (ANOVA) with Tukey's post hoc for comparison between treatments. However, if the data show anormal distribution, Friedman to compare the different times in the same group (intra group), and Kruskal Wallis to make the comparison between groups (inter group). To evaluate the QEHD ordinal data, Wilcoxon and Mann-Whitney tests will be used. Bioestat 5.3 (Belém, Pará, Brazil) will be used, considering an alpha level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Two to four hypersensitive teeth with a response ≥ 04 on the visual analogue scale (VAS) from 0 to 10, where 0 represents no pain and 10 extreme pain, during the application of tactile (explorer probe) and evaporative (jet air);
* Dentinal exposure on the posterior teeth, due to the presence of a shallow non-carious lesion up to 02 mm in depth, according to the Smith & Knight index (measured with a millimeter probe), and / or class I gingival recession according to Miller classification.

Exclusion Criteria:

* Restorations; tooth decay and/or periodontal pockets; dental pulpitis; enamel cracks or fractures on sensitive teeth;
* Continuous treatment with anti-inflammatory drugs and/or analgesics or desensitizing treatment induced three months prior to research recruitment data;
* Pregnancy or lactation;
* Systemic diseases;
* Fixed orthodontic appliances;
* Occlusal instability.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Dentin hypersensitivity | 30 days
  The evaluation of dentin hypersensitivity will be performed with three (3) evaluation times: baseline (immediately before the beginning of treatment), 15 and 30 days, through tactile and evaporative stimuli, using the visual analog scale (VAS) from 0 to 10, where 0 represents no pain and 10 extreme pain.

SECONDARY OUTCOMES:
Quality of life | 30 days
  The self-reported evaluation of the volunteers will be completed through a questionnaire before the beginning and after one month with the completion of the research to determine the impact of treatment on their quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Cecy M Silva, PhD, Study Chair — Federal University of Pará
Locations (1):
- Universidade Federal do Pará, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: No